CLINICAL TRIAL: NCT00007384
Title: Longitudinal LDL-C Studies in Black and White Families
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 957; R01HL062394 (NIH)
Record Dates: First submitted 2000-12-19; First posted 2000-12-19 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2008-01

CONDITIONS: Cardiovascular Diseases; Atherosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis

SUMMARY:
To longitudinally investigate multigenerational familial clustering of plasma low density lipoprotein cholesterol (LDL-C), with particular emphasis on the influences of apoE genotypes and various 'behaviors'.

DETAILED DESCRIPTION:
BACKGROUND:

Elevated concentrations of plasma low density lipoprotein cholesterol (LDL-C), a major risk factor for coronary heart disease, cluster significantly in families. This clustering has been observed in cross-sectional studies in both black and white families, but longitudinal data on the familial clustering of LDL-C are virtually nonexistent.

DESIGN NARRATIVE:

The longitudinal study will provide new and important information about changes in the familial low density lipoprotein cholesterol (LDL-C) correlations in black and white families from the period of shared household environments to that of separate households, using families from the Princeton Lipid Research Clinics (LRC) Prevalence (1973-75) and Family Studies (1975-76). The study will also provide important information on changes in individual LDL-C levels over the same 25 year period. The former student participants were six to 18 years of age and are now 32 to 45 years of age; their parents were (largely) 26 to 55 years of age and are now 51 to 80 years of age. Plasma LDL-C concentrations in children and adults have been shown to associate with the apolipoprotein (apo) E genotype, with obesity, and with such elective behaviors as diet, cigarette smoking, and physical activity. In the LRC Study, measurements were made of LDL-C, body habitus, elective behaviors, and the family history of cardiovascular disease (CVD). The study will obtain repeat measures of these factors, plus determine the apo E isoforms. Changes in individual LDL-C levels and in familial associations can then be assessed in association with apo E isoforms, body composition, elective behaviors, and family history of CVD. Family members share ranges of body weight, patterns of fat distribution, dietary and smoking habits, and physical activity levels. The extent to which the familial clustering of LDL-C levels is determined by apo E isoforms interacting with the similar levels of obesity, and with the similar behaviors, is not currently known.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-07; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Morrison — Children's Hospital & Medical Center

REFERENCES:
- [Background] Miles MV, Horn PS, Tang PH, Morrison JA, Miles L, DeGrauw T, Pesce AJ. Age-related changes in plasma coenzyme Q10 concentrations and redox state in apparently healthy children and adults. Clin Chim Acta. 2004 Sep;347(1-2):139-44. doi: 10.1016/j.cccn.2004.04.003. PMID 15313151
- [Background] Miles MV, Morrison JA, Horn PS, Tang PH, Pesce AJ. Coenzyme Q10 changes are associated with metabolic syndrome. Clin Chim Acta. 2004 Jun;344(1-2):173-9. doi: 10.1016/j.cccn.2004.02.016. PMID 15149886
- [Background] Miles MV, Horn PS, Morrison JA, Tang PH, DeGrauw T, Pesce AJ. Plasma coenzyme Q10 reference intervals, but not redox status, are affected by gender and race in self-reported healthy adults. Clin Chim Acta. 2003 Jun;332(1-2):123-32. doi: 10.1016/s0009-8981(03)00137-2. PMID 12763289